CLINICAL TRIAL: NCT03328065
Title: Viewpoints on the Social Representations and Rationale Concerning the Choices of Patients, Doctors and Caregivers With Regard to the Management of Patients With Non-resectable Metastatic Cancer of the Colon, Stomach, Bile Ducts, Rectum, Pancreas or Lung, or Gastrointestinal Neuroendocrine Tumours
Acronym: EOLE
Status: Terminated | Type: Observational
Why Stopped: lack of inclusion
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: LEJEUNE FdF 2016
Record Dates: First submitted 2017-10-04; First posted 2017-11-01 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Non-resectable Metastatic Cancer of the Lung; Non-resectable Metastatic Cancer of the Colon; Non-resectable Metastatic Cancer of the Rectosigmoid Junction; Non-resectable Metastatic Cancer of the Stomach; Non-resectable Metastatic Cancer of the Bile Duct; Non-resectable Metastatic Cancer of the Rectum; Non-resectable Metastatic Cancer of Gastrointestinal Neuroendocrine Tumour; Non-resecable Metastatic Cancer of the Pancreas
MeSH Terms: interventions — Interviews as Topic; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Stable patients, early responders to treatment and caregivers
  Interventions: Other: Interviews; Other: Questionnaires
- Stable patients and intermediate responders and c: Stable patients and intermediate responders to treatments and caregivers
  Interventions: Other: Interviews; Other: Questionnaires
- Doctors
  Interventions: Other: Interviews; Other: Questionnaires
- Patients in therapeutic escape and their caregivers
  Interventions: Other: Interviews; Other: Questionnaires

INTERVENTIONS:
Other: Interviews — Semi-directed interviews, recorded and transcribed for analysis
Other: Questionnaires — economic and psycho-social questionnaires

SUMMARY:
Reflexion on the therapeutic strategies to implement in patients at the end of life is advancing rapidly in France. However, beyond the choices presented to patients, sometimes even the decision to carry on, to limit or to stop treatments is also questioned. This decision is subjective; it is influenced by the patient's representation system (emotions, beliefs, values, practices, etc). In addition, even though he or she is the focus of the decision, the patient is not alone; other actors, accompanying the patient, play an important role in the final decision making. These actors, namely the doctors and close relatives, are also influenced in their decision making. This coexistence of representation systems may interfere with objective indicators that help in decision making (functional, clinical and biological) or with the knowledge acquired by doctors in their training and may complicate the decision-making process.

ELIGIBILITY:
Inclusion Criteria:

I- PATIENTS

* men or women
* who have been informed about the study
* and who have provided verbal consent to take part in the study
* able to understand written and spoken French
* with non-resectable metastatic cancer of: the colon, or the rectosigmoid junction or the stomach or bile ducts or rectum or gastrointestinal neuroendocrine tumor or lung (not small-cell cancer) or pancreas
* with a caregiver designated as the principal caregiver (family, friend, neighbour)
* who has consented to the principal caregiver taking part in a qualitative interview
* able to take part in an interview lasting roughly one hour

II- CAREGIVERS

* men or women
* who have been informed about the study
* who have provided verbal consent to take part in the study
* able to understand written and spoken French
* able to follow an interview lasting roughly one hour

III-DOCTORS

* men or women
* who have been informed about the study
* who have provided verbal consent to take part in the study
* specialised in specific organ or oncologist prescriber

Exclusion Criteria:

I- PATIENTS

* under guardianship or ward of court
* with a severe handicap (neurological disease: Parkinson, Alzheimer, other dementia, multiple sclerosis, severe mental retardation etc.)

II- CAREGIVERS

* under guardianship or ward of court,
* with a severe handicap (neurological disease: Parkinson, Alzheimer, other dementia, multiple sclerosis…),
* with severe mental retardation impairing ability to understand.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: hospitalized patients
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2017-12-19 (Actual); Primary Completion 2020-12-09 (Actual); Study Completion 2020-12-19 (Actual)

PRIMARY OUTCOMES:
Number of determinants which are privileged by the patients to choose a treatment | through study completion, an average of 18 months
Type of determinants which are privileged by the patients to choose a treatment | through study completion, an average of 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourogne, Dijon, France